CLINICAL TRIAL: NCT06740110
Title: A Histomorphometric Analysis of Bone Formation With Two Different Bone Graft Material in Adult Patients Required Socket Preservation After Tooth Extraction
Brief Title: Bone Material's Histomorphometric Analysis In Socket Preservation
Acronym: BM-HIS-SP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Inventi S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC-MD-CIP-003
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-06

CONDITIONS: Socket Preservation
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): The intervention will include tooth extraction and GBR procedure. After clinical and radiographic assessment, local anaesthesia is applied. The dentist performs atraumatic extraction, cleans the socket, places investigational device, and applies gauze for hemostasis. The patient is given post-operative care instructions. After recovery the first and second stage of implantation will be performed.
  Interventions: Device: Tooth extraction and GBR procedure
- Standard of care arm (Active Comparator): The intervention will include tooth extraction and GBR procedure. After clinical and radiographic assessment, local anaesthesia is applied. The dentist performs atraumatic extraction, cleans the socket, places standard of care device and applies gauze for hemostasis. The patient is given post-operative care instructions. After recovery the first and second stage of implantation will be performed.
  Interventions: Device: Tooth extraction and GBR procedure

INTERVENTIONS:
Device: Tooth extraction and GBR procedure — The intervention will include tooth extraction and GBR procedure. After clinical and radiographic assessment, local anaesthesia is applied. The dentist performs atraumatic extraction, cleans the socket, places investigational device (first arm) or standard of care (second arm) and applies gauze for hemostasis. The patient is given post-operative care instructions. After recovery the first and second stage of implantation will be performed.

SUMMARY:
This is a prospective, multicentre, parallel-group, randomized controlled, single blinded (participant) trial aims to compare the investigational medical device with standard of care in dental treatment addressing the preservation of bone loss after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with full legal capacity, male and female;
* Patients with ability to understand the proposed surgical treatment and to understand and sign the informed consent;
* Patients who are willing and able to comply with scheduled visits, treatment and other trial procedures;
* Patients who respect the follow-up recalls.

Exclusion Criteria:

* Presence of bone lesions;
* Patients with alcohol or substance abuse;
* Patients with smoking habits (more than 10 cigarettes per day);
* Patients presenting physical and/or mental handicap that impede an adequate oral hygiene;
* Pregnant or breast feeding women;
* Patients currently participating in any other clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quantify the new bone formation via histomorphometric analysis following tooth extraction with GBR procedure. | 6 months
  A new bone formation assesses via histomorphometric evaluation.

SECONDARY OUTCOMES:
Evaluation of (serious) adverse events (S)AEs. | 13 months
  Number of (S)AEs

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Indywidualna Praktyka Stomatologiczna Marek Śmielecki, Gniezno
  - Medicare, Mińsk Mazowiecki
  - Stomatologia Niteckie Sp. z o.o., Tychy
  - Rafał Dobrakowski Dentysta, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided